CLINICAL TRIAL: NCT07040488
Title: Study of Infrared Thermography in Diabetic Foot in Guadeloupe (ETPDG)
Brief Title: Study of Infrared Thermography in Diabetic Foot in Guadeloupe
Acronym: ETPDG
Status: Recruiting | Type: Observational
Sponsor: Centre Hospitalier Universitaire de la Guadeloupe (Other)
Responsible Party: Sponsor
Other Study IDs: PAP_RIPH2_2024/03; 2024-A00993-44 (Other: ANSM Frech Human Health Organisation)
Record Dates: First submitted 2025-06-11; First posted 2025-06-27 (Actual); Last update posted 2025-06-27 (Actual); Status verified 2025-06

CONDITIONS: Diabetic Foot Infection
Keywords: Infrared thermography; diabetic foot; infection
MeSH Terms: conditions — Diabetic Foot; Infections

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- non-diabetic individuals (control group): Healthy volunteers will be recruited from the post-emergency consultation service of the ambulatory medicine platform at CHUG. These are patients attending for a follow-up evaluation after a previous visit to the emergency department.
- diabetic individuals with diabetic foot ulceration: Diabetic patients with foot ulceration will be recruited during their visits to the multidisciplinary consultation at the Diabetic Foot Unit of the University Hospital of Guadeloupe, or during their hospitalizations in the orthopedic surgery department.
- diabetic individuals without diabetic foot ulceration: Diabetic patients without foot ulceration will be recruited from the diabetes day hospital at CHUG, the ambulatory medicine platform at CHUG, and the diabetes therapeutic education program.

SUMMARY:
It is hypothesized that thermal imaging differs between diabetic and non-diabetic individuals in Guadeloupe. Infrared thermography is also suggested as a useful tool for studying diabetic foot ulceration. The main objective is to compare the temperatures of four areas of the plantar surface of the foot among non-diabetic individuals, diabetic individuals, and diabetic individuals with foot ulceration.

DETAILED DESCRIPTION:
Diabetes represents a major public health issue in the region. Among its most severe complications is diabetic foot ulceration, which frequently results in amputation. Infrared thermography is a non-invasive and non-ionizing imaging technique that provides precise temperature data at specific points on the body. When combined with 3D imaging technologies, infrared thermography may offer early diagnostic potential for infections related to diabetic foot ulcers, by revealing both visible and subclinical signs. A preliminary step in assessing the relevance of thermal imaging is to determine whether thermographic patterns differ between the feet of diabetic and non-diabetic individuals within the Guadeloupean population, particularly in a tropical climate. Currently, international guidelines do not recommend infrared thermography as part of routine clinical practice for managing diabetic foot ulceration. However, this imaging modality could potentially contribute to the diagnostic arsenal for infections associated with diabetic foot ulcers.

ELIGIBILITY:
Inclusion Criteria for Control Group

* Adult patients
* Patients of Afro-Caribbean origin
* Volunteer patients free from pathology
* Person affiliated to or beneficiary of a social security scheme.
* Person who has agreed to sign a consent to participate in the study

Inclusion Criteria for diabetic patients:

* Adult patients
* Patients of Afro-Caribbean origin
* Type 1 or type 2 diabetic patients with and without diabetic foot ulceration
* Person affiliated to or beneficiary of a social security system.
* Person who has agreed to sign a consent to participate in the study

Exclusion Criteria :

* - Minors
* patient with an active fracture or a history of fracture
* a history of legs surgery
* History of amputation
* Bilateral diabetic ulceration
* neurological disease (Parkinson, stroke, etc.)
* pregnancy
* Foot mycosis
* refusal of consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy volunteers will be recruited from the post-emergency consultation service of the ambulatory medicine platform at CHUG. These are patients attending for a follow-up evaluation after a previous visit to the emergency department.
  Diabetic patients without foot ulceration will be recruited from the diabetes day hospital at CHUG, the ambulatory medicine platform at CHUG, and the diabetes therapeutic education program.
  Diabetic patients with diabetic foot ulceration will be recruited during their visits to the multidisciplinary consultation at the Diabetic Foot Unit of the University Hospital of Guadeloupe or during their hospitalizations in the orthopedic surgery department. Based on data from previous years, the active patient list consulting the Diabetic Foot Unit (UPPD) for foot ulceration is estimated to exceed 300 individuals.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2024-09-27 (Actual); Primary Completion 2026-03-27 (Estimated); Study Completion 2026-03-27 (Estimated)

PRIMARY OUTCOMES:
temperatures at four areas of the plantar surface of the foot | baseline
  The primary outcome is the measurement of temperatures in degrees Celsius (°C) using infrared thermography (coupled with a 3D camera) at four areas of the plantar surface of the foot: the pulp of the hallux, the heel, the heads of the first and fifth metatarsals, and at the site of the diabetic foot ulcer.

SECONDARY OUTCOMES:
Temperatures on the same area of the contralateral foot | baseline
  Temperatures in degrees Celsius (°C) at the level of the ulceration of the diabetic foot and on the same area of the contralateral foot

CONTACTS AND LOCATIONS:
Overall Officials: Vanéva CHINGAN-MARTINO, MD, Principal Investigator — CHU de la Guadeloupe
Locations (1):
- Chu de La Guadeloupe, Pointe-à-Pitre, Guadeloupe

IPD SHARING:
Plan to Share IPD: Undecided